CLINICAL TRIAL: NCT04094402
Title: Epi-GERD Study: Epidemiological Evaluation in Patients With Gastro-Esophageal Reflux
Brief Title: Epi-GERD Study: Epidemiological Evaluation in Patients With Gastro-Esophageal Reflux Disease (GERD)
Acronym: Epi-ERGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scandinavia Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: Epi-ERGE
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None. It is an observational study — None. It is an observational study

SUMMARY:
Cross-sectional epidemiological study in patients with diagnosis of GERD (Gastroesophageal Reflux Disease) and with current treatment or with a history of recent treatment with some PPI (Proton Pump Inhibitor), in order to evaluate the persistence and / or relapse of symptoms of GERD.

DETAILED DESCRIPTION:
OBJECTIVE: To carry out an evaluation about the persistence and / or relapse of symptoms in Colombian patients with diagnosis of GERD.

MATERIALS AND METHODS: A multicentric cross-sectional epidemiological study will be carried out in Colombian patients with diagnosis of GERD and with current treatment or with a history of recent treatment with some PPI (Proton Pump Inhibitor). The persistence and / or relapse of symptoms will be evaluated as the main variable. The secondary variables to be evaluated include: Demographical analysis, treatment (s) used by patients, adverse events associated with the treatments, comorbidities and risk factors. The analysis will be carried out from two perspectives: A first descriptive approach and a second analytical approach, with a level of significance of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Previous diagnosis of Gastroesophageal Reflux Disease (GERD)
* CURRENT treatment with a proton-pump inhibitor (PPI), OR NOT CURRENT treatment with some PPI but YES in the last year

Exclusion Criteria:

* Refusal to participate in the study by the patient.
* Patients who, in the judgment of the Investigator, do not understand or are not willing to adequately answer to the questions.
* Mental or psychiatric illness that, in the judgment of the investigator, does not allow adequate information to be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years, with previous diagnosis of Gastroesophageal Reflux Disease (GERD)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Symptoms of GERD (Gastroesophageal Reflux Disease) | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years
  Proportion of patients with persistence and / or relapse of symptoms of GERD.

SECONDARY OUTCOMES:
Demographic analysis | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years
  Characterization of patients
Kind of IBP taked by the patient and the way to consume it. | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years
  A descriptive analysis of the type of IBP types taken by patients and how to take them
Adverse Events related with the treatments | It will be evaluated in each patient (only once, at the time of the interview) throughout the study which is estimated to last 3 years
  Evaluation of Adverse events associated with the treatment (s)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Castillo, Dr, Study Director — Medical Director
Locations (1):
- Scandinavia Pharma, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No